CLINICAL TRIAL: NCT02554435
Title: TAME Health: Testing Activity Monitors' Effect on Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-0014
Record Dates: First submitted 2015-08-24; First posted 2015-09-18 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity
Keywords: physical activity; activity monitor; older adults; 5 A's counseling
MeSH Terms: conditions — Motor Activity

ARMS (2):
- Pedometer (Active Comparator): All participants will be given 5 A's counseling and a digital pedometer (Digi-walker CW-700/701, YAMAX, San Antonio, TX). Participants will be asked to log their daily steps measured by the pedometer in an activity diary.
  Interventions: Behavioral: 5 A's counseling; Device: Pedometer
- Electronic Activity Monitor (EAM) (Experimental): All participants will be given an EAM (UP24 by Jawbone, San Francisco, CA) and the corresponding UP24 application (app) on their smart device. In addition to monitoring activity, the app allows for social comparison and social interaction. Participants will "friend" other participants to utilize these features.
  Interventions: Device: EAM; Behavioral: 5 A's counseling

INTERVENTIONS:
Device: EAM — The monitor provides the participant feedback on their daily steps, active time, idle time, burned calories, and distance traveled through the mobile application (app). Participants can review all of their feedback while in the intervention. If the participants chose, they are also able to monitor their sleep and dietary intake. The app also provides health tips and daily challenges. The participants will also have the opportunity to interact with other participants through the social features of the app.
  Other Names: UP24; Jawbone; Electronic Activity Monitor
  Arms: Electronic Activity Monitor (EAM)
Behavioral: 5 A's counseling — Brief counseling to encourage behavioral change. The counseling is intended to be administered by a health care provider. The component of the counseling are assess, advise, agree, assist, and arrange.
Device: Pedometer — The pedometer provides the participant feedback on their daily steps, activity time, distance traveled, and calories burned. Participants can review the feedback for the past 7 days.
  Arms: Pedometer

SUMMARY:
Cardiovascular disease accounts for 1 in 3 deaths among US adults and is strongly related to physical activity. Most older adults do not participate in healthy levels of physical activity. Physical activity promotion and counseling from a primary health care provider is important for disease prevention. In addition to counseling, an activity monitor can increase physical activity through self-regulation. Two types of monitors are available: pedometers and electronic activity monitors (EAMs). Research shows that both monitors are motivational devices that can increase physical activity. Pedometers count steps of the wearer. EAMs can monitor steps, monitor burned calories, quality of sleep, and sedentary time. EAMs may also offer more behavioral change techniques and opportunities for self-monitoring. The goal of this study is to compare the effectiveness of EAMs compared to a pedometer on increasing physical activity and decreasing cardiovascular risk within older adult, primary care patients. The study will include sedentary, overweight primary care patients, 55-74 years of age with access to a smart phone or tablet. All participants will receive brief physical activity counseling. Participants will then be randomized to receive a self-monitoring device (Digi-walker CW-700/701 or UP24 by Jawbone) to wear for 3 months. Investigators will evaluate the following outcomes: physical activity, cardiovascular risk (Framingham risk calculator, fitness), psychological feeling toward exercise, physical function, health status, exercise motivation and self-regulation. The investigators hypothesize that EAMs will be more effective than pedometers in improving these outcomes. The results of this pilot test will aid in the translation of effective physical activity intervention components to primary care clinics for cardiovascular disease prevention.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is prevalent and the leading cause for mortality in the United States. The American Heart Association's (AHA) 2020 Impact Goal is to improve the cardiovascular health of all Americans by 20 percent while reducing deaths from CVD and stroke by 20 percent. Maintaining healthy levels of physical activity (PA) is critical in maintaining cardiovascular health, but older adults are inactive. Inactivity may be influenced by low levels of motivation. Standard behavioral counseling techniques typically implemented within the primary care setting target increased motivation, but lack the key component of self-control. The addition of electronic activity monitors (EAMs) that provide interactive self-monitoring, feedback, and social support may further increase motivation for exercise by providing more effective behavior change techniques than standard protocols. Investigators will conduct a three month intervention trial that will test the feasibility of adding an EAM system to brief counseling within a primary care setting. Participants (N = 40) will be randomized to receive evidence-based brief counseling plus either an EAM or a pedometer. Investigators propose two Specific Aims:

AIM 1: Evaluate the feasibility and acceptability of implementing a technology-enhanced brief intervention to increase physical activity in a primary care setting. Measures of feasibility will include days the EAM was worn, usage of the app, technological problems, attrition, and adverse events. Acceptability will be measured by self-report and focus groups.

AIM 2: Compare the counseling plus EAM intervention to a counseling plus pedometer intervention. Primary outcomes will be changes in PA and cardiovascular risk. We will also investigate secondary outcomes (differences in adherence, weight and body composition, health status, motivation, physical function, psychological feelings, self-regulation).

ELIGIBILITY:
Inclusion Criteria:

* physically inactive (less than 60 minutes per week)
* BMI between 25-35
* in good health measured by Par-Q+
* access to a smart phone

Exclusion Criteria:

* physical activity is inadvisable by their doctor
* involved in another physical activity intervention within the past 6 months
* used an activity monitor in the past 6 months
* unwilling to travel for scheduled visits
* currently taking medications that affect body composition
* current smoker
* report alcohol or drug problem
* institutionalized for psychiatric illness within the last year
* do not consent

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zakkoyya Lewis, BS, Principal Investigator — The University of Texas Medical Branch
Locations (2):
- United States (2):
  - Primary Care Pavilion, Galveston, Texas
  - Victory Lakes Town Center, League City, Texas

REFERENCES:
- [Background] Lewis ZH, Ottenbacher KJ, Fisher SR, Jennings K, Brown AF, Swartz MC, Lyons EJ. Testing Activity Monitors' Effect on Health: Study Protocol for a Randomized Controlled Trial Among Older Primary Care Patients. JMIR Res Protoc. 2016 Apr 29;5(2):e59. doi: 10.2196/resprot.5454. PMID 27129602
- [Derived] Lewis ZH, Ottenbacher KJ, Fisher SR, Jennings K, Brown AF, Swartz MC, Martinez E, Lyons EJ. Effect of Electronic Activity Monitors and Pedometers on Health: Results from the TAME Health Pilot Randomized Pragmatic Trial. Int J Environ Res Public Health. 2020 Sep 18;17(18):6800. doi: 10.3390/ijerph17186800. PMID 32961834
- [Derived] Lewis ZH, Ottenbacher KJ, Fisher SR, Jennings K, Brown AF, Swartz MC, Martinez E, Lyons EJ. The feasibility and RE-AIM evaluation of the TAME health pilot study. Int J Behav Nutr Phys Act. 2017 Aug 14;14(1):106. doi: 10.1186/s12966-017-0560-5. PMID 28807041
- See also: TAME health protocol citation — http://www.researchprotocols.org/2016/2/e59/

RESULTS

PARTICIPANT FLOW:
Groups:
- Electronic Activity Monitor: All participants will be given an EAM (UP24 by Jawbone, San Francisco, CA) and the corresponding UP24 application (app) on their smart device. In addition to monitoring activity, the app allows for social comparison and social interaction. Participants will "friend" other participants to utilize these features.
  EAM: The monitor provides the participant feedback on their daily steps, active time, idle time, burned calories, and distance traveled through the mobile application (app). Participants can review all of their feedback while in the intervention. The app also provides health tips and daily challenges. The participants will also have the opportunity to interact with other participants through the social features of the app.
  5 A's counseling: Brief counseling to encourage behavioral change. The counseling is intended to be administered by a health care provider. The component of the counseling are assess, advise, agree, assist, and arrange.
Period: Overall Study
Arm/Group | Pedometer | Electronic Activity Monitor
Started | 20 | 20
Completed | 14 | 19
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pedometer | Electronic Activity Monitor | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (5.7) | 64.0 (5.1) | 63.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 2 | 3 | 5
  Black/African-American | 3 | 4 | 7
  Other | 1 | 1 | 2
  Non-Hispanic White | 14 | 12 | 26
Physical Activity [Mean (Standard Deviation); unit: minutes per day] — Physical activity was defined as the minutes of moderate to vigorous physical activity as measured by the Sensewear Armband.
  minutes per day | 40.0 (33.9) | 22.5 (21.5) | 31.3 (29.4)
Steps [Mean (Standard Deviation); unit: steps per day] | 4560.18 (2285.6) | 3849.4 (2107.8) | 4204.8 (2199.8)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Minutes Measured by a SenseWear Armband
Description: Minutes of moderate-vigorous physical activity over a 7 day period
Time Frame: Physical activity minutes at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
minutes per day | 40.2 (3.7) | 33.8 (27.6)

2. Primary Outcome: Composite Measure for Cardiovascular Risk Measured by the Framingham Non-laboratory Risk Calculator
Description: Factors within the risk calculator include of age in years, systolic blood pressure, gender, and body mass index. These factors are used to create a composite score to estimate the individual's risk for a cardiac event within the next 10 years. The risk score is not bound by maximums and minimums, however a lower number is more favorable. Among women, a composite risk score of 10 equates to a 6% risk of a cardiovascular event, a risk score of 15 equates to a 13% risk, a risk score of 20 equates to a 28.5% risk, and a risk score of 21 or higher equates to >30% risk of a cardiovascular event within the next 10 years. Among men, a composite risk score of 10 equates to a 9% risk, a risk score of 15 equates to a 21.5% risk, and a risk score of 18 or higher equates to >30% risk of a cardiovascular event within the next 10 years.
Time Frame: Cardiovascular risk at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: Risk score
Groups:
- Electronic Activity Monitor: All participants will be given an EAM (UP24 by Jawbone, San Francisco, CA) and the corresponding UP24 application (app) on their smart device. In addition to monitoring activity, the app allows for social comparison and social interaction. Participants will "friend" other participants to utilize these features.
  EAM: The monitor provides the participant feedback on their daily steps, active time, idle time, burned calories, and distance traveled through the mobile application (app). Participants can review all of their feedback while in the intervention. If the participants chose, they are also able to monitor their sleep and dietary intake. The app also provides health tips and daily challenges. The participants will also have the opportunity to interact with other participants through the social features of the app.
  5 A's counseling: Brief counseling to encourage behavioral change. The counseling is intended to be administered by a health care provider. The component of the
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
Risk score | 21.2 (12.6) | 16.6 (13.2)

3. Primary Outcome: 6-minute Walk Test
Description: distance walked in 6 minutes
Time Frame: Fitness at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
feet | 1642.9 (287.3) | 1561 (353.6)

4. Primary Outcome: Steps Per Day
Description: Measured by a SenseWear Armband. Average steps per day over a 7 day period
Time Frame: Steps per day at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
steps | 4702 (2259.7) | 4353 (2021.4)

5. Secondary Outcome: Weight
Time Frame: Weight at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
kg | 86.8 (13.6) | 81.9 (11.2)

6. Secondary Outcome: Body Mass Index (BMI)
Time Frame: BMI at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
kg/m^2 | 30.5 (3.1) | 30.0 (3.5)

7. Secondary Outcome: Waist-to-Hip Ratio
Description: Waist-to-Hip ratio was calculated by divided the waist circumference (in inches) by the hip circumference (in inches).
Time Frame: Waist-to-hip ratio at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
ratio | .84 (0.1) | 0.80 (0.1)

8. Secondary Outcome: Blood Pressure
Time Frame: Blood pressure at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
mmHg
  Systolic blood pressure | 134.3 (14.6) | 125.0 (14.5)
  Diastolic blood pressure | 83.4 (10.0) | 80 (9.8)

9. Secondary Outcome: Exercise Motivation
Description: Measured by Behavioral Regulation in Exercise Questionnaire-2. Sub-scales include intrinsic, identified, introjected, extrinsic, and amotivation. Each subscale ranges from 0 - 4, with 0 being lowest and 4 being highest level of motivation for the given subscale. The different subscales measure varying forms of autonomous motivation; therefore high scores (maximum of 4) of "intrinsic" and "identified" are better. Alternatively, low scores of "introjected", "extrinsic", and "amotivation" are better.
Time Frame: Exercise motivation at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
units on a scale
  Intrinsic | 1.48 (1.0) | 2.84 (0.77)
  Identified | 2.24 (1.04) | 2.92 (0.59)
  Introjected | 1.12 (1.06) | 1.68 (0.88)
  Extrinsic | 0.49 (0.69) | 0.51 (0.58)
  Amotivation | 0.61 (0.78) | 0.15 (0.38)

10. Secondary Outcome: Quality of Life Measured by the SF-36 Questionnaire
Description: Sub-scales include physical functioning, social functioning, physical role limitations, emotional role limitations, mental health, energy/vitality, and pain. All sub-scales have a range of 0 to 100. High scores and scores closer to 100 represent a better outcome for each sub-scale.
Time Frame: Quality of life at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
units on a scale
  Physical functioning | 62.3 (29.3) | 73.1 (19.3)
  Social functioning | 75.8 (25.5) | 71.3 (31.4)
  Physical role limitations | 67.9 (26.6) | 72.2 (24.2)
  Emotional role limitations | 75.8 (25.5) | 71.3 (31.4)
  Mental health | 70 (18.6) | 76.3 (18.7)
  Energy/vitality | 53.1 (15.1) | 58.1 (16.7)
  Pain | 56.8 (29.1) | 60.3 (26.1)

11. Secondary Outcome: Physical Function Measured by the Short Physical Performance Battery
Description: Physical function is operationalized by 3 functional tests, including repeated chair stands (5 consecutive stands), balance (semi-tandem stand, side-by-side stand, tandem stand) and 8 feet walk. The time it took for participants to complete each test was timed in seconds. The faster the repeated chair stand and 8 feet walk tests were performed, the better the function of the individual. Therefore, lower scores represent a better outcome. These tests were not bound by maximums. The higher score for tandem balance, maximum of 10, represents a better outcome. The balance test is comprised of three positions but time is only recorded for one. Participants start with the semi-tandem, then if they are able to hold the position for 10 seconds they continue to tandem balance test. If they are not able to hold the semi-tandem position for 10 seconds, they then complete the side by side test. In this study, all participants proceeded to the tandem test, so outcome is labeled "tandem balance."
Time Frame: Physical function at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
seconds
  Chair stand | 14.2 (3.7) | 14.7 (5.5)
  Tandem balance | 9.2 (2.2) | 9.1 (2.4)
  8 feet up and go | 5.9 (1.4) | 6.4 (3.0)

12. Secondary Outcome: Psychological Feelings
Description: Measured by the Psychological Need Satisfaction in Exercise Scale. Sub-scales include perceived competence, perceived autonomy, and perceived relatedness. Each sub-scale had a range from 1 to 5. Higher scores, in each sub-scale, represent a more favorable outcome.
Time Frame: Psychological feelings at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
units on a scale
  Competence | 2.49 (0.94) | 3.43 (0.95)
  Autonomy | 3.16 (0.95) | 4.01 (0.95)
  Relatedness | 2.72 (1.33) | 3.53 (1.03)

13. Secondary Outcome: Resting Pulse
Time Frame: Resting pulse at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
bpm | 76.5 (11.9) | 69.1 (14)

14. Secondary Outcome: Change From Baseline in Self-regulation
Description: Measured by the Rovinak et al scale. Sub-scales include exercise goals and exercise plans. The possible scores on both subscales range between 10 and 50, with higher scores representing more favorable outcomes in exercise goals and planning.
Time Frame: Change in self-regulation from baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pedometer | Electronic Activity Monitor
Number analyzed (Participants) | 20 | 20
units on a scale
  Goal-setting | 22.1 (5.3) | 31.3 (9.8)
  Planning | 24.3 (4.1) | 26.4 (7.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Pedometer | Electronic Activity Monitor
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pedometer (N=20) | Electronic Activity Monitor (N=20)
Knee replacement (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Two participants had knee replacement surgery after consenting to the study, but their participation in the study did not start until they completed physical therapy.
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant was admitted to the hospital for kidney stones
Adverse reaction (Product Issues) | 1 (1) | 0 (0) — Participant had an adverse reaction to physician prescribed medication for a chronic illness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No